CLINICAL TRIAL: NCT00219232
Title: An Open-label Extension to Evaluate the Efficacy and Safety of the Rivastigmine Transdermal Patch in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713D2320E1
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

INTERVENTIONS:
Drug: Rivastigmine Transdermal Patch

SUMMARY:
The goal of this research study is to evaluate, in the open-label extension phase, the safety and efficacy of the rivastigmine transdermal patch in patients with probable Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled the inclusion and exclusion criteria as listed in the study CENA713D2320 and have completed the double-blind treatment phase on study medication without significant protocol violations.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2003-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by adverse events, vital signs and skin irritation for up to 28 weeks treatment

SECONDARY OUTCOMES:
Change in cognition from baseline (week 24 of the double blind phase) at week 52
Clinical global impression of change from baseline at week 52
Change in activities of daily living from baseline at week 52
Change in behavioral symptoms from baseline at week 52
Change in executive function from baseline at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Result] Grossberg G, Sadowsky C, Frostl H, Frolich L, Nagel J, Tekin S, Zechner S, Ros J, Orgogozo JM. Safety and tolerability of the rivastigmine patch: results of a 28-week open-label extension. Alzheimer Dis Assoc Disord. 2009 Apr-Jun;23(2):158-64. doi: 10.1097/wad.0b013e31818b1c2c. PMID 19484917